CLINICAL TRIAL: NCT06296667
Title: Effect of Core Muscles Training On Patients With Chronic Mechanical Low Back Pain According To SALIBA'S Postural Classification System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Saleh Elemam Yassin, researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003644
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- group1: vertical/ vertical (Experimental): participant posture: The thoracic block is vertically aligned over the pelvic block.The angle of the thoracic block is vertical in the sagittal plane allowing for the dome of the diaphragm to rest on top of the abdomen.Vertical force transfers through the musculoskeletal system through the mid-foot and into the standing surface causing no shifts in postural alignment.
  Interventions: Other: core muscles training exercises
- group 2: vertical/ posterior (Experimental): participant posture: The thoracic block is vertically aligned over the pelvic block but is posteriorly tipped in the sagittal plane.Vertical force leads to an accentuated extension in the thoracolumbar and lumbar regions with decreased ability to sustain vertical forces.
  Interventions: Other: core muscles training exercises
- group 3: posterior/ posterior (Experimental): participant posture: The thoracic block is aligned posterior to the pelvic block and is posteriorly tipped in the sagittal plane. Vertical force leads to an accentuated extension in the lower lumbar region with a forward shear of the pelvis and decreased ability to sustain vertical forces.
  Interventions: Other: core muscles training exercises
- group 4: posterior/ anterior (Experimental): participant posture: The thoracic block is aligned posterior to the pelvic block and is anteriorly tipped in the sagittal plane. Vertical force leads to a slight flexion in the thoracic and lumbar regions with a forward shear of the pelvis and decreased ability to sustain vertical force.
  Interventions: Other: core muscles training exercises
- group 5:anterior/ posterior (Experimental): participant posture: The thoracic block is aligned anterior to the pelvic block and is posteriorly tipped in the sagittal plane. Vertical force leads to extension in the mid and lower lumbar regions with a posterior shear of the pelvis and decreased ability to sustain vertical forces.
  Interventions: Other: core muscles training exercises
- group 6: anterior/ anterior (Experimental): participant posture: The thoracic block is aligned anterior to the pelvic block and is anteriorly tipped in the sagittal plane. Vertical force leads to an overall flexion of the trunk and decreased ability to sustain vertical forces
  Interventions: Other: core muscles training exercises

INTERVENTIONS:
Other: core muscles training exercises — The sessions will be conducted three times per week for four weeks and each exercise will be performed two sets of 10 repetitions. For the static exercises, the final position will be held for 6 second. There will be a pause of 3 second between repetitions, and a 60 sec rest between each exercise. The exercise will be performed in three forms: abdominal bracing, dynamic stabilization, and advanced core strengthening.

SUMMARY:
This study is designed as a pre and post experimental study. The purposes of this study are to evaluate the effect of core muscles training in patients with chronic mechanical low back pain according to SALIBA'S postural classification system (SPCS) in terms of pain intensity, function, and core muscles endurance.

DETAILED DESCRIPTION:
Male and female patients diagnosed with chronic mechanical low back pain will be referred to physical therapy department. Patients will then be screened based on the inclusion and exclusion criteria of the current study. They will be asked to sign the informed consent form. Then, participants will be assessed for the severity of pain, functional disability, and core endurance test at baseline and at the end of the treatment by the same physiotherapist.

In addition, participants will be instructed to stand in habitual posture while looking forward and will be photographed from sagittal plane wearing shorts(males) and a thin clothes(female). The photos will be used to subjectively classify the patients into one of the 6 postural classification groups (G1, G2, G3,G4, G5, G6). The Vertical compression test and elbow flexion test will be used to objectively confirm the classification.

Later, photos will be then entered by researcher to Kinovea software for more objective confirmation of the classification.

Then, Participants will be allocated purposive randomly to one of the six groups according to evaluation criteria(saliba's postural classification system).

Then, Patients in each postural category will receive a 4-week program of core muscles training.

Two tests will be used to further confirm the classification of patients' posture.

These tests are:

1. Vertical compression test (VCT): Patient position: the patient will be asked to stand in a natural position and relax everything but the knees (so as not to buckle and collapse when pressure is applied) Therapist's position and manual contact: Standing side by side or stride position, therapist may be positioned on a stool, chair, or table. Therapist positions forearms vertical then hovers and place hands on the patient's shoulders, between the acromion and the first rib insertion. Therapist must ensure that all force is directed to patient and not allow movement in his or her body unless patient buckles. Therapist's action and verbal command: After instruction, apply gentle, sustained pressure vertically through the patient's trunk or pelvis. Gradually build the pressure from a grade of (1) which is at the point. Where the therapist feels the pressure of the patient's bony surfaces through the soft tissue covering the carpal ridge, to a (2) which is double the pressure of (1), and then to a (3) which is triplethe pressure of (1), and so on until full force is applied which would be a grade of (5). An efficient response is one in which the pressure applied by the therapist translates evenly to the base of support. In standing that would be to the arch of the foot, translating into the second ray. An efficient response is a springy end feel An inefficient response (failure) is noted when the pressure applied by the therapist causes the spine to side bend, backward bend, shear or rotate. In addition, an inefficient response is a hard end feel.

2-Elbow flexion test (EFT): Purpose: to test the proper timing of core and global muscles in response to an external load through the forearms and confirm findings of the CoreFirst Patient's position: In Standing, patient's elbows will be bent to 90 degrees, forearms supinated to loose-packed position and humerus is perpendicular to the floor, not flexed or extended and no substitution of shoulder adduction allowed to assist in stabilization. Therapist's position and manual contact: Therapist stands in front of patient, may be in squat position for resistance from below and therapist may also apply resistance from above. Therapist positions forearms perpendicular to floor then hovers. Hand placement is over the distal end of the forearm. Verbal command: "Don't let me straighten your arms". Once the command is given, the therapist gradually increases the downward resistance, being cautious NOT to pull forward while pushing or pulling down. Grading is 1-5, with "1" defined as the amount of pressure requires to feel the bones of your hands on the bones of the patient's forearms, and 2 = 2x1, 3 = 3x1, 4 = 4x1, and 5 - 5x1. When applying the resistance, the therapist asks the patient to note where the effort is and how hard it feels to maintain the position. The patient should note if the effort is in the cervical, shoulder girdle, thoracic spine, lumbar spine, or forearms. An efficient state is one in which the patient can maintain the elbow position through automatic activation of the core, rotator cuff, shoulder girdle, and global shoulder and arm muscles. The spine should remain stable, and the patient should maintain his balance. In an inefficient state, the patient will attempt to maintain the position with global muscles and will often give in the arms, shoulder girdle, and spine. The patient will frequently fall forward as the force is applied or tilt the upper body back to compensate for the load.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred with a diagnosis of CMLBP of at least 3 months.

  * Age ranging from 20 to 55 years old.
  * Both genders will be included.
  * BMI(18.5-24.9).

Exclusion Criteria:

* Lumbar canal stenosis.

  * History of vertebral fractures.
  * patients with neurological deficits such as altered sensation.
  * Spinal surgery or failed back surgery.
  * cardiovascular/ pulmonary disorder

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
pain intensity. | one month
  Pain intensity will be assessed using the visual analog scale (VAS). The VAS is a unidimensional measure of pain intensity. It is a continuous scale comprises of a horizontal line 10 cm in length. The scale is anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10). A higher score indicates greater pain intensity
function disability | one month
  Functional disability will be estimated using the cross-culturally adapted Arabic version of the Oswestry disability questionnaire.The score is calculated by the addition of the values assigned for each of the 10 individual questions and is used to categorize disability as: mild or no disability (0- 20%); moderate disability (21%-40%); severe disability (41% to 60%); incapacity (61% to 80%); restricted to bed (81% to 100%).
core muscles endurance | one month
  The researcher will conduct a series of core stability tests before and after the core training program. The following core tests will be used: trunk flexion test (McGill's test) , Trunk extension (Sorenson Test, Right Side plank test,left side plank and prone plank test. We will record the time (in seconds) the patient can hold the isometric posture, with a normal range of 1-2 minutes

OTHER OUTCOMES:
participants gender will be male and females, their age in years,their height in meters,weight in kilograms. | one month
  ( weight and height will be combined to report body mass index (BMI) (e.g., weight divides on height^2 in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University,Faculty of Physical Therapy, Giza, Egypt